CLINICAL TRIAL: NCT04842344
Title: A Prospective Randomized Controlled Trial of Extracorporeal Carbon Dioxide Removal (ECCO2R) in the Treatment of Acute Exacerbation of Chronic Obstructive Pulmonary Disease With Severe Hypercapnia
Brief Title: ECCO2R in the Treatment of Acute Exacerbation of COPD With Severe Hypercapnia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Li Xuyan (Other)
Responsible Party: Sponsor-Investigator, Li Xuyan, Sponsor Investigator, Beijing Chao Yang Hospital
Organization: Beijing Chao Yang Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2020-KE-492
Record Dates: First submitted 2021-04-08; First posted 2021-04-13 (Actual); Last update posted 2021-04-13 (Actual); Status verified 2021-04

CONDITIONS: Lung Diseases, Obstructive
Keywords: Acute exacerbation of chronic obstructive pulmonary disease; extracorporeal carbon dioxide removal; Hypercapnia respiratory failure
MeSH Terms: conditions — Lung Diseases, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Noninvasive ventilation and ECCO2R (Experimental)
  Interventions: Device: ECCO2R
- Noninvasive ventilation (No Intervention)

INTERVENTIONS:
Device: ECCO2R — extracorporeal carbon dioxide removal
  Arms: Noninvasive ventilation and ECCO2R

SUMMARY:
Patients with moderate to severe acute exacerbation of chronic obstructive pulmonary disease are often complicated with hypercapnia and respiratory failure, so they need to be admitted to ICU for monitoring and respiratory support treatment. Noninvasive ventilation has become the first-line respiratory support for the treatment of AECOPD with hypercapnia and respiratory failure. However, 26-54% of AECOPD patients with hypercapnia and respiratory failure eventually fail to receive noninvasive ventilation and need endotracheal intubation and invasive ventilation to maintain effective gas exchange. For these patients, the in-hospital survival rate is only 31-76%, and the prognosis is poor. In AECOPD patients with high risk of noninvasive ventilation failure and expected need of intubation, timely giving other ways of respiratory support to reduce blood CO2 may avoid patients receiving tracheal intubation and invasive ventilation, thus avoiding related complications and adverse prognosis. As a new type of respiratory support technology, ECCO2R is worthy of attention in monitoring and evaluation of support effect in AECOPD patients with respiratory failure. It is urgent that ECCO2R can effectively alleviate respiratory failure, avoid complications related to tracheal intubation, improve quality of life and reduce mortality.

ELIGIBILITY:
Inclusion Criteria:

* AECOPD patients.
* The patients with hypercapnia respiratory failure were admitted to ICU and needed noninvasive ventilation.
* The results of blood gas analysis showed pH <7.30, PaCO2> 50 mmHg.
* There were high risk factors for failure of noninvasive ventilation: after receiving continuous 2 hours of noninvasive ventilation, the arterial blood pressure showed the pH value was ≤ 7.30, while PaCO2 was 20% higher than the baseline value, and any one or more of the following conditions were combined: respiratory rate ≥ 30 times / min, assisted respiratory muscle breathing; contradictory breathing.
* Informed consents were sighed.

Exclusion Criteria:

* The mean arterial pressure was less than 60 mmHg after volume and vasoactive drug treatment.
* There were anticoagulant contraindications.
* Weight over 120kg.
* Patients with malignant tumor or other complications, the expected survival time was less than 30 days.
* It could not cooperate with noninvasive ventilation or has contraindication of noninvasive ventilation.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 176 (Estimated)
Dates: Start 2021-05-01 (Estimated); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-03-31 (Estimated)

PRIMARY OUTCOMES:
Demand rate of endotracheal intubation | 28 days

SECONDARY OUTCOMES:
Actual rate of endotracheal intubation | 28 days
hospital mortality | 28 days
length of ICU stay | 28 days
length of hospital stay | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Bing Sun, MD, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Institute of Respiratory Medicine, Beijing Chao-yang Hospital, Capital Medical University, Beijing, China